CLINICAL TRIAL: NCT04009317
Title: A Multicenter, Randomized, Open-label Study to Evaluate the Efficacy and Safety of TQ-B3139 Versus Crizotinib in the First Line Treatment of Subjects With Anaplastic Lymphoma Kinase (ALK) Positive Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study of TQ-B3139 Versus Crizotinib in the First Line Treatment of Subjects With Anaplastic Lymphoma Kinase (ALK) Positive Non-Small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3139-III-01
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-07

CONDITIONS: ALK-positive NSCLC
MeSH Terms: interventions — Crizotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQ-B3139 (Experimental): TQ-B3139 tablet 600mg administered orally , twice daily in 28-day cycle.
  Interventions: Drug: TQ-B3139
- Crizotinib (Active Comparator): Crizotinib tablet 250mg administered orally, twice daily in 28-day cycle.
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: TQ-B3139 — a multi-target protein kinase inhibitor.
  Arms: TQ-B3139
Drug: Crizotinib — a multi-target protein kinase inhibitor.
  Arms: Crizotinib

SUMMARY:
To evaluate the efficacy and safety of TQ-B3139 versus crizotinib in subjects with ALK-positive NSCLC that have received one chemotherapy regimen and have not received ALK inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* 1.18 and 75 years. 2. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.

  3. Life expectancy ≥12 weeks. 4. Histologically or cytologically confirmed advanced or metastatic NSCLC with ALK-positive.

  5. Has not received ALK tyrosine kinase inhibitor (TKI). 6. Has received one chemotherapy regimen for stage IIIB-IV NSCLC. 7. At least one measurable lesion. 8. Adequate organ system function. 9. Understood and signed an informed consent form.

Exclusion Criteria:

* 1. Has diagnosed and/or treated additional malignancy within 5 years prior to randomization. Exceptions include cured cancer carcinoma in situ of the cervix, intramucosal carcinoma of gastrointestinal tract, breast and melanoma skin cancers and superficial bladder tumors.

  2. Hypersensitivity to TQ-B3139 or crizotinib. 3. Has received any cancer therapy within 4 weeks or 5 times of t1/2. 4. Has received any major surgery within 4 weeks. 5. Has received any radiotherapy or minor surgery aimed to cure cancer within 2 weeks.

  6. Acute toxicity that is ≥ Grade 2 caused by previous cancer therapy. 7. Has active viral, bacterial and fungal infections within 2 weeks before the first dose.

  8. Has serious cardiovascular disease within 3 months before the first dose. 9. Has currently uncontrollable congestive heart failure. 10. Has continuous arrhythmia ≥ Grade 2, uncontrollable atrial fibrillation or QTc interval > 480ms.

  11. Has interstitial fibrosis or interstitial lung disease ≥ Grade 3. 12. Brain metastases with symptom. 13. HBsAg positive and HBV DNA positive (≥ULN);HCV antibody and HCV-RNA positive (≥ULN); HIV positive or ≥HIV ULN.

  14. Has multiple factors affecting oral medication. 15. Has received a strong CYP3A inhibitors within 7days before the first dose. 16. Has received a strong CYP3A inducers. 17. Breastfeeding or pregnant women.; Men unwilling to use adequate contraceptive measures during the study.

  18. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2019-08-13 (Actual); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | up to 36 months
  PFS defined as the time from randomization until the first documented progressive disease (PD) or death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 36 months
  Percentage of subjects achieving complete response (CR) and partial response (PR).
Disease Control rate (DCR) | up to 36 months
  Percentage of subjects achieving CR, PR, stable disease (SD) and Non-CR/Non-progressive disease (PD)
Overall Survival (OS) | up to 36 months
  OS defined as the time from randomization to death from any cause. Subjects who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Yang Y, Min J, Yang N, Yu Q, Cheng Y, Zhao Y, Li M, Chen H, Ren S, Zhou J, Zhuang W, Qin X, Cao L, Yu Y, Zhang J, He J, Feng J, Yu H, Zhang L, Fang W. Envonalkib versus crizotinib for treatment-naive ALK-positive non-small cell lung cancer: a randomized, multicenter, open-label, phase III trial. Signal Transduct Target Ther. 2023 Aug 14;8(1):301. doi: 10.1038/s41392-023-01538-w. PMID 37574511